CLINICAL TRIAL: NCT00445341
Title: A Phase I/II Study of Flavopiridol in Relapsed or Refractory Mantle Cell Lymphoma (MCL) and Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Flavopiridol to Treat Relapsed Mantle Cell Lymphoma or Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Roschewski, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070081; 07-C-0081
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Lymphoma
Keywords: Microarray; Proteomics; Hybrid Schedule; Tumor Lysis Syndrome; Cyclin D1; Lymphoma; Mantle Cell Lymphoma; MCL; Diffuse Large B-Cell Lymphoma; DLBCL
MeSH Terms: conditions — Lymphoma; Tumor Lysis Syndrome; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — alvocidib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Flavopiridol in lymphoma patients (Experimental): Flavopiridol 30 mg/m^2 is given weekly for 4 weeks followed by a 2 week break for up to 6 cycles. It is given through a vein as a 30 minute infusion followed by a 4 hour infusion.
  Interventions: Drug: Flavopiridol

INTERVENTIONS:
Drug: Flavopiridol — Flavopiridol 30 mg/m^2 is given weekly for 4 weeks followed by a 2 week break for up to 6 cycles. It is given through a vein as a 30 minute infusion followed by a 4 hour infusion.
  Other Names: alvocidib

SUMMARY:
Background:

Mantle cell lymphoma (MCL) and diffuse large B-cell lymphoma (DLBCL) are aggressive subtypes of non-Hodgkin lymphoma.

Flavopiridol is an investigational drug that works differently from standard chemotherapy and may target abnormalities in MCL and DLBCL cells, such as a protein excess that prevents tumor cells from dying.

A challenge in developing flavopiridol for treatment has been determining its optimal dosing schedule. The schedule used for this study is effective in a type of leukemia called chronic lymphocytic leukemia (CLL) and may benefit patients with MCL and DLBCL also.

Objectives:

To determine the highest dose of flavopiridol that can be given safely to patients with relapsed MCL and DLBCL at the dosing schedule detailed below

To assess the response of the tumor to flavopiridol given at the test dosing schedule

Eligibility:

Patients 18 years of age and older with relapsed MCL or DLBCL

Design:

Flavopiridol is given at four different dose levels, starting with the lowest dose for the first group of three to six patients and increasing with subsequent groups, depending on side effects at the preceding dose. The drug is given weekly for 4 weeks followed by a 2-week break (one cycle) for up to six cycles. It is given through a vein as a 30-minute infusion followed by a 4-hour infusion.

Patients undergo the following procedures for research studies and to evaluate the effect of treatment on the tumor:

* Blood tests
* Lymph node, bone marrow and tumor biopsies
* Lymphapheresis to collect blood cells for research
* Disease staging with imaging studies (computed tomography (CT), positron emission tomography (PET) and/or magnetic resonance imaging (MRI) after every 2 cycles

DETAILED DESCRIPTION:
Background:

Flavopiridol is a synthetic N-methylpiperidinyl, chlorophenyl flavone compound that targets a number of different cellular pathways and processes.

It works through several different mechanisms that include inhibition of cyclin dependent kinases and the cyclin D-1 complex which is over-expressed in mantle cell lymphoma. Flavopiridol also has demonstrated activity in activated B-like diffuse large B-cell lymphoma cell lines.

One of the great challenges in developing flavopiridol and applying it clinically has been determining its optimal dosing schedule. Following several different dosing schedules, one strategy that has been very promising in chronic lymphocytic leukemia (CLL) is the application of so-called hybrid schedules of the drug (an infusion for an intermediate time following a bolus dose).

Objectives:

Assess the toxicity and safety of administration of this hybrid schedule.

Assess the response rate of the hybrid schedule of flavopiridol in relapsed mantle cell lymphoma (MCL) and diffuse large B-cell lymphoma (DLBCL).

Eligibility:

Relapsed MCL or DLBCL.

Eastern Cooperative Oncology Group (ECOG) performance status(P.S.) less than or equal to 2.

Age greater than or equal to 18 years.

Human immunodeficiency virus (HIV) serology negative

Design:

Phase I/II.

Phase I portion consists of 3-4 dose levels of 3-6 patients each.

Administer weekly times 4 and then 2 weeks off (1 cycle). Restage after every 2 cycles. Continue if complete response (CR), partial response (PR) or stable disease (SD) for up to 6 cycles. Dose reductions for toxicity will be addressed in the protocol.

Phase II portion of the study will be a Simon optimal two-stage design: designed to rule out 20% response rate (p0=0.20) in favor of a 45% response rate (p1=0.45).

The maximum sample size to be accrued for this study will be 71 patients.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Previously treated mantle cell lymphoma or diffuse large B-cell lymphoma (to include mediastinal (thymic) large B-cell lymphoma; transformed large B-cell lymphoma; follicular grade IIIB large B-cell lymphoma; intravascular large B-cell lymphoma).

Confirmed pathological diagnosis at the National Cancer Institute, National Institutes of Health (NIH).

Recurrent measurable disease (measurable disease in 2 dimensions or leukemic disease which can be quantified and followed).

Prior anthracycline-based treatment for patients with diffuse large B-cell lymphoma (DLBCL).

Age greater than 18 years.

Eastern Cooperative Oncology Group (ECOG) performance 2 or better.

Major organ function: absolute neutrophil count (ANC) greater than 1000/mcL, Platelet greater than 50,000/mcL, Creatinine less than 1.5 mg/dL or creatinine clearance greater than 60 mL/min; serum glutamic pyruvic transaminase (SGPT) less than 5 x upper limit of normal; bilirubin less than 2 mg/dL (total) except less than 5 mg/dL in patients with Gilbert's syndrome as defined by greater than 80% unconjugated. ANC and platelet requirements must be met independent of transfusion.

Informed consent and willingness to use contraception by both men and women.

Both male and female patients must be willing to use adequate contraception (to include effective barrier methods of contraception) or to completely abstain from heterosexual intercourse while on protocol treatment.

EXCLUSION CRITERIA:

Pregnant or nursing because of an unknown potential for teratogenic or abortifacient effects.

Human immunodeficiency virus (HIV) serology negative. HIV positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with flavopiridol. Additionally, the biology of HIV associated DLBCL's is often quite different from HIV negative disease due to involvement of Epstein Barr virus (EBV).

Hepatitis B surface antigen negative.

Active central nervous system (CNS) lymphoma. These patients have a poor prognosis and because they frequently develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse events.

History of inflammatory bowel disease unless this has been inactive for a period of 2 or more years.

Recovery from toxicity of prior therapy to a grade 1 or less.

Systemic cytotoxic or experimental treatments within 4 weeks of treatment.

White blood cell (WBC) greater than 100,000 cells/mcL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-11-27 (Actual); Primary Completion 2012-04-30 (Actual); Study Completion 2012-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Roschewski, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Worland PJ, Kaur G, Stetler-Stevenson M, Sebers S, Sartor O, Sausville EA. Alteration of the phosphorylation state of p34cdc2 kinase by the flavone L86-8275 in breast carcinoma cells. Correlation with decreased H1 kinase activity. Biochem Pharmacol. 1993 Nov 17;46(10):1831-40. doi: 10.1016/0006-2952(93)90590-s. PMID 8250970
- [Background] Arguello F, Alexander M, Sterry JA, Tudor G, Smith EM, Kalavar NT, Greene JF Jr, Koss W, Morgan CD, Stinson SF, Siford TJ, Alvord WG, Klabansky RL, Sausville EA. Flavopiridol induces apoptosis of normal lymphoid cells, causes immunosuppression, and has potent antitumor activity In vivo against human leukemia and lymphoma xenografts. Blood. 1998 Apr 1;91(7):2482-90. PMID 9516149
- [Background] Byrd JC, Peterson BL, Gabrilove J, Odenike OM, Grever MR, Rai K, Larson RA; Cancer and Leukemia Group B. Treatment of relapsed chronic lymphocytic leukemia by 72-hour continuous infusion or 1-hour bolus infusion of flavopiridol: results from Cancer and Leukemia Group B study 19805. Clin Cancer Res. 2005 Jun 1;11(11):4176-81. doi: 10.1158/1078-0432.CCR-04-2276. PMID 15930354
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-C-0081.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flavopiridol in Lymphoma Patients
Started | 28
Completed | 26
Not Completed | 2
Not completed — refused further treatment | 1
Not completed — taken off treatment too early | 1

BASELINE CHARACTERISTICS:
Arm/Group | Flavopiridol in Lymphoma Patients
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.71 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (e.g. Toxicity)
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 47 months
Measure: Count of Participants; unit: Participants
Arm/Group | Flavopiridol in Lymphoma Patients
Number analyzed (Participants) | 28
Participants | 28

2. Primary Outcome: Response Rate (Complete Response (CR) and Partial Response (PR))
Description: Response was assessed by the Cheson criteria. Complete response is complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease related symptoms if present before therapy, and normalization of those biochemical abnormalities (e.g.(LDH) definitely assignable to the lymphoma. All lymph nodes must have regressed to normal size (</= 1.5 cm in greatest diameter if > 1.5 cm before therapy). Previously involved nodes that were 1.1 to 1.5 cm in greatest diameter must have decreased to </= 1 cm or by more than 75% in the sum of the products of the greatest diameters (SPD). Spleen, if considered to be enlarged before therapy, must have regressed in size. Partial response is a >/= 50% decrease in the SPD of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease. Splenic and hepatic nodules must regress by >/= 50% in the SPD. Bone marrow is irrelevant for determination of a PR.
Time Frame: 2/16/2007 - 1/20/2011
Measure: Count of Participants; unit: Participants
Arm/Group | Flavopiridol in Lymphoma Patients
Number analyzed (Participants) | 26
Participants
  Complete Response | 0
  Partial Response | 2

ADVERSE EVENTS:
Time Frame: 47 months
Arm/Group | Flavopiridol in Lymphoma Patients
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 14/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flavopiridol in Lymphoma Patients (N=28)
Cardiac troponin I (cTnI) (Cardiac disorders) | 1 (1)
Conduction abnormality/atrioventricular heart block::AV Block-Third degree (Complete AV block) (Cardiac disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema: head and neck (Blood and lymphatic system disorders) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 2 (2)
Hypotension (Cardiac disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L::Colon
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Abdomen NOS (Reproductive system and breast disorders) | 1 (1)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 2 (3)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 2 (2)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 3 (3)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flavopiridol in Lymphoma Patients (N=28)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 13 (47)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 22 (84)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 23 (136)
Alkaline phosphatase (Metabolism and nutrition disorders) | 16 (33)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 8 (8)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 9 (13)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 12 (31)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 4 (6)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 4 (15)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 9 (23)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 9 (15)
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 22 (99)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema: limb (Blood and lymphatic system disorders) | 6 (6)
Edema: trunk/genital (Blood and lymphatic system disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9 (11)
Febrile neutropenia (Infections and infestations) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >= 38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 7 (9)
Glomerular filtration rate (Metabolism and nutrition disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6 (12)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 22 (145)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Cardiac disorders) | 7 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Urinary tract NOS
Infection with normal ANC or Grade 1 or 2 neutrophils::Bladder (urinary) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Colon (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Pharynx (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Rectum (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 1 (1)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 24 (148)
Lymphopenia (Blood and lymphatic system disorders) | 26 (156)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 12 (30)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 16 (61)
Mood alteration::Depression (Nervous system disorders) | 1 (1)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 2 (2)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal/Soft Tissue - Other (Specify, calf cramping) (Musculoskeletal and connective tissue disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 25 (48)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 22 (108)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 6 (8)
Pain::Abdomen NOS (Reproductive system and breast disorders) | 3 (3)
Pain::Back (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain::Head/headache (Nervous system disorders) | 2 (2)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 2 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 19 (79)
Platelets (Blood and lymphatic system disorders) | 21 (112)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 7 (15)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 8 (25)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Rigors/chills (General disorders) | 2 (2)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 8 (25)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 16 (37)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 2 (2)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (2)
Syncope (fainting) (Nervous system disorders) | 3 (4)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 5 (13)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 2 (2)
Vision-blurred vision (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 16 (40)
Weight gain (General disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2011-06-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT00445341/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-10-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT00445341/Prot_SAP_001.pdf